CLINICAL TRIAL: NCT03548480
Title: Targeting the Gut Microbiome for Prader-Willi Syndrome Treatment
Acronym: BALPWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FSJD-BALPWS-2018
Record Dates: First submitted 2018-05-02; First posted 2018-06-07 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Placebo — Intervention with a daily dose of placebo
  Arms: Placebo
Dietary Supplement: Probiotic — Intervention with a daily dose of probiotic
  Arms: Probiotic

SUMMARY:
The gut microbiome has recently emerged as a major contributor to obesity, systemic inflammation, and metabolic disease. Furthermore, intestinal bacteria are crucial players in the gut-brain axis, regulating a broad range of central nervous system processes, from satiety mechanisms to anxiety and social behavior. Thus, targeting the microbiome is being actively investigated as a therapeutic strategy for a wide array of diseases, including obesity, anxiety, depression, and autism. Among all intestinal bacteria, Bifidobacterium animalis spp. lactis (BAL) has shown promise for obesity treatment in experimental animal models and human subjects, improving body composition and metabolic health, and reducing energy intake. Moreover, tryptophan metabolism, a crucial regulator of satiety mechanisms and anxiety, is a main target of BAL. Given that clinical manifestations of Prader-Willi syndrome (PWS) include hyperphagia, anxiety, altered body composition, and metabolic dysregulation, the aforementioned effects of BAL might prove highly beneficial for children with PWS. Here, the investigators will test this hypothesis by performing a randomized double-blinded placebo-controlled crossover clinical study to assess the effects of BAL supplementation on an array of clinical manifestations of PWS. Children with PWS will undergo a 3-month placebo/probiotic treatment period, a 3-month washout period, followed by a 3-month probiotic/placebo supplementation. Anthropometric, biochemical, and psychological data as well as biological samples will be obtained at the beginning of the study, and after each of the study periods, with a total of four time-points. Specifically, the investigators will determine body composition by DXA analysis; metabolic health by assessing glucose and lipid metabolic parameters as well as circulating hormonal and cytokine levels; thermoregulation by non-invasive thermal imaging; and hyperphagia and emotional and behavioral problems by applying parental-rated validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Prader-Willi Syndrome with genetic confirmation
* On a stable diet and medication regimen for at least the last two months before enrollment

Exclusion Criteria:

* Current enrollment in or discontinuation within the last 30 days from a clinical trial
* Presence of other medical problems that would preclude study participation
* Patients with a history of bariatric surgery
* Unsuitable for inclusion in the study in the opinion of the investigator

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in percent body fat | 3 months
  Measured by DXA scan

SECONDARY OUTCOMES:
Change in lipid profile (triglyceride, cholesterol) | 3 months
  Blood test after overnight fasting
Change in glucose metabolic parameters (glucose, insulin, HbA1c) | 3 months
  Blood test after overnight fasting
Change in circulating cytokine levels | 3 months
  Quantified in plasma samples
Change in hyperphagia | 3 months
  Measured by validated questionnaire (HQ-CT)
Change in thermoregulation | 3 months
  Measured by thermal imaging

OTHER OUTCOMES:
Change in plasma metabolome | 3 months
  Liquid chromatography coupled to mass spectrometry will be used to obtain a comprehensive metabolic profile of plasma samples
Change in urine metabolome | 3 months
  Liquid chromatography coupled to mass spectrometry will be used to obtain a comprehensive metabolic profile of urine samples
Change in intestinal microbiome | 3 months
  DNA isolated from fecal samples will be analyzed by sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Carles Lerin, PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amat-Bou M, Garcia-Ribera S, Climent E, Piquer-Garcia I, Corripio R, Sanchez-Infantes D, Villalta L, Elias M, Jimenez-Chillaron JC, Chenoll E, Ramon D, Ibanez L, Ramon-Krauel M, Lerin C. Effects of Bifidobacterium animalis Subsp. lactis (BPL1) Supplementation in Children and Adolescents with Prader-Willi Syndrome: A Randomized Crossover Trial. Nutrients. 2020 Oct 13;12(10):3123. doi: 10.3390/nu12103123. PMID 33066107